CLINICAL TRIAL: NCT06154460
Title: Comparison of Different Surgical Stabilization Methods for Recurrent Anterior Shoulder Instability in Terms of Pain, Proprioceptive Sense, Functional Status, and Muscle Activation
Brief Title: The Effects of Different Surgical Stabilization Methods in Recurrent Anterior Shoulder Instability
Acronym: SSM-SI
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Ferruh Taşpınar, Study Director, Izmir Democracy University
Other Study IDs: SSM-SI-35
Record Dates: First submitted 2023-11-02; First posted 2023-12-04 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Surgery; Anterior Shoulder Instability
Keywords: Joint Instability; Shoulder Joint; Orthopedic Procedurs; Shoulder Pain; Proprioception; Functional Status; Electromyography
MeSH Terms: conditions — Joint Instability; Shoulder Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Laterjet Surgery Group: This group will consist of individuals who underwent laterjet surgery.
  Interventions: Procedure: Laterjet Surgery
- Reimplissage Surgery Group: This group will consist of individuals who underwent reimplissage surgery.
  Interventions: Procedure: Reimplissage Surgery
- Capsular Reconstruction Surgery Group: This group will consist of individuals who underwent capsular reconstruction surgery.
  Interventions: Procedure: Capsular Reconstruction

INTERVENTIONS:
Procedure: Laterjet Surgery — The laterjet procedure is an operation in which the coracoid process is transferred to the glenoid rim with a screw.
  Other Names: LS
  Groups: Laterjet Surgery Group
Procedure: Reimplissage Surgery — Reimplissagge operation, which means "to fill", is an open procedure designed to limit the engagement of Hill-Sachs deformity by passing the infraspinatus into the Hill-Sachs defect.
  Other Names: RS
  Groups: Reimplissage Surgery Group
Procedure: Capsular Reconstruction — Allografts or autografts are used for capsular reconstruction. In the procedure performed with capsular repair and grafts, the capsule is strengthened and stabilization is attempted
  Other Names: CR
  Groups: Capsular Reconstruction Surgery Group

SUMMARY:
Shoulder instability is the inability to retain the humeral head in the glenoid fossa. The incidence of instability is 8.2 to 23.9 per 100,000 person-years with an estimated prevalence of 1.7%. The most common shoulder instability with a rate of 98% is anterior dislocation, in which the humeral head is displaced anterior to the glenoid. Conservative and surgical treatments of instability are available. There are many controversial issues related to these methods in the literature. For example; an atrophy and functional loss in the infraspinatus after reimplissage, atrophy and loss of proprioception in the muscles around the shoulder after capsular repair, and loss of proprioception after the laterjet procedure have been reported.Therefore, the aim of this study was to compare different surgical stabilization methods in terms of pain, proprioceptive sensation, functional status and muscle activation in recurrent anterior shoulder instability, which is very common in adults.

DETAILED DESCRIPTION:
Shoulder instability is the inability to retain the humeral head in the glenoid fossa. The incidence of instability is 8.2 to 23.9 per 100,000 person-years with an estimated prevalence of 1.7%. The most common shoulder instability with a rate of 98% is anterior dislocation, in which the humeral head is displaced anterior to the glenoid. It is more common in young males. While damage is limited to the capsule and labrum in most instabilities seen in young people, rotator cuff tear is also observed in 89% of those over 40 years of age. Trauma is the main cause of shoulder instability. While 96% of shoulder instabilities develop as a result of a blow to the arm in abduction or external rotation of the shoulder with excessive flexion, approximately 4% occur without trauma. Anterior instability occurs when the shoulder is forced into abduction and external rotation by impact, and posterior instability occurs when the shoulder in slight flexion and adduction is hit. The glenohumeral joint is an unstable joint because the depth and size of the glenoid fossa are not fully compatible with the humerus and as a result, the range of motion is wider compared to other joints in the body. While articular surface congruence, articular version, glenoid labrum, capsule and ligaments constitute static factors in ensuring stability; rotator cuff, biceps tendon, intra-articular negative pressure and muscles that form scapulothoracic movements (Trapezoid, Serratus Anterior, Rhomboids, Latissimus Dorsi) constitute dynamic factors. Insufficiency of one or more of these structures causes instability. Conservative and surgical treatments of instability are available. Conservative treatment includes nonoperative methods. These methods consist of electrophysical agents, heat-light agents, exercise and manual treatment methods and proceed through a certain protocol according to the patient's condition and symptoms. In cases where medical and physical therapies are not sufficient, surgical treatment procedures are initiated.

Reimplisasagge, capsular reconstruction and laterjet methods are commonly used in surgical treatments. Reimplissagge operation, which means "to fill", is an open procedure designed to limit the engagement of Hill-Sachs deformity by passing the infraspinatus into the Hill-Sachs defect. The possibility of loss of internal and external rotation as a result of infraspinatus tendon transfer after reimplissage is a matter of debate. Allografts or autografts are used for capsular reconstruction, which is another surgical method. In the procedure performed with capsular repair and grafts, the capsule is strengthened and stabilization is attempted. The laterjet procedure is an operation in which the coracoid process is transferred to the glenoid rim with a screw.

There are many controversial issues related to these methods in the literature. For example; an atrophy and functional loss in the infraspinatus after reimplissage, atrophy and loss of proprioception in the muscles around the shoulder after capsular repair, and loss of proprioception after the laterjet procedure have been reported. Therefore, the aim of our study was to compare these commonly applied methods in terms of pain, proprioceptive sensation, functional status and muscle activation and the hypothesis of the study was as follows; Hypothesis of the Study: Laterjet, reimplissage and capsular reconstruction surgical procedures in recurrent anterior shoulder instabilities affect pain, proprioceptive sensation, functional status and muscle activation differently.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* At least 4 months after surgery,
* Not having any diagnosed neurological problem

Exclusion Criteria:

* Having an additional diagnosis that would cast doubt on the assessments (rheumatoid arthritis, cancer, neurological disorders, fibromyalgia, psychiatric disorders, etc.),
* Pregnancy status or suspicion
* Having undergone a different surgery such as a fracture with instability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample of the study will consist of individuals who have undergone surgery in the Department of Orthopedics and Traumatology of Dokuz Eylül University Hospital due to instability diagnosis and who have returned to their activities of daily living. The research groups will consist of 30 patients with at least 10 patients each for 3 different surgical methods. These methods will be compared with each other in terms of pain, proprioceptive sensation, functional status and muscle activation. According to the reviewed studies, the number of individuals to be included in the study was determined as 30 individuals in total, 10 in each group.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | Subjects will be evaluated between a post-operative minimum of 4 months and a maximum of 2 years.
  Pain will be assessed by visual analog scale (VAS). A 10 cm horizontal line will be used for this. '0' means no pain and '10' means the worst possible pain
Assessment of proprioceptive sensation | Subjects will be evaluated between a post-operative minimum of 4 months and a maximum of 2 years.
  Positioning test will be used for the evaluation of proprioceptive sensation. Evaluation scores are calculated as the proportion of correct responses for repositioning.
Assessment of Range of Motion | Subjects will be evaluated between a post-operative minimum of 4 months and a maximum of 2 years.
  A universal goniometer will be used for normal range of motion assessment. The normal limits of active range of motion are considered to be 180° for shoulder flexion, 180° for shoulder abduction, 90° for shoulder external rotation and 70-90° for shoulder internal rotation.
Assessment of Hand Grip Strength | Subjects will be evaluated between a post-operative minimum of 4 months and a maximum of 2 years.
  Hand grip strength will be assessed with jamar hand dynamometer. In the test procedure, 3 measurements are made for hand grip and finger grip strengths with one-minute intervals between each measurement and the averages are recorded. High values mean high grip strength.
Assessment of functional status | Subjects will be evaluated between a post-operative minimum of 4 months and a maximum of 2 years.
  DASH (Disability Arm Shoulder and Hand) questionnaire will be used. Each item has 5 response options ranging from 'no difficulty or no symptoms' to 'unable to perform the activity or very severe symptom' and is scored on a scale of 1 to 5 points. A scale score ranging from 0 (no disability) to 100 (most severe disability) is calculated.
Assessment of Shoulder Instability | Subjects will be evaluated between a post-operative minimum of 4 months and a maximum of 2 years.
  WOSI (Western Ontario Shoulder Instability Index) will be used. The WOSI is a 21-item questionnaire used for patients with shoulder instability. Each question results in a number between 0 and 100 and the total score is presented as a number between 0 and 2100 points.
Assessment of Muscle Activation | Subjects will be evaluated between a post-operative minimum of 4 months and a maximum of 2 years.
  Muscle activation will be evaluated by superficial EMG measurements. For this, the muscles with the best reaction around the shoulder joint were selected. These muscles were musculus infraspinatus, musculus middle deltoideus, musculus upper trapezius and musculus pectoralis major. The activation of the muscles will be evaluated during isometric contraction and during isotonic contractions performed in 3 different planes and results will be interpreted according to activation status. Data will be recorded during maximum voluntary isometric contraction (MVIC) and isotonic contraction (IC). During these contacts, the calculated "area" on the chart will be recorded. Additionally, the "IC/MVIC" percentage will be calculated to determine the workload on the muscle during the activity.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Özkan, Prof. Dr., Principal Investigator — Dokuz Eylul University; Betul Taspinar, Prof. Dr., Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No